CLINICAL TRIAL: NCT01223664
Title: The Efficacy of Allogenic Bone Marrow Stem Cells Transplantation in Patients With Liver Cirrhosis Resulting From Chronic Hepatitis B
Brief Title: Allogenic Bone Marrow Stem Cells Transplantation in Patients With Liver Cirrhosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Lin Bingliang, Third Affiliated Hospital, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYS-1012
Record Dates: First submitted 2010-10-12; First posted 2010-10-19 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Liver Cirrhosis
Keywords: ABMSC; Allogenic bone marrow mesenchymal stem cells; Liver cirrhosis; Transplantation
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A(conserved therapy ) (Active Comparator): Thirty of the enrolled patients were assigned to Group A were received comprehensive treatment including antiviral drugs, lowering aminotransferase and jaundice medicine.
  Interventions: Drug: Conserved therapy
- Group B (BMSC Transplantion) (Experimental): Thirty of the enrolled patients were assigned to Group B to receive comprehensive treatment including antiviral drugs, lowering aminotransferase and jaundice medicine, as well as bone marrow stem cells transplantation
  Interventions: Procedure: Allogenic bone marrow stem cells transplantation

INTERVENTIONS:
Procedure: Allogenic bone marrow stem cells transplantation — 30ml allogenic bone marrow stem cells were infused to patients using interventional method via portal vein or hepatic artery as well as conserved therapy
  Arms: Group B (BMSC Transplantion)
Drug: Conserved therapy — Oral or intravenous administration
  Arms: Group A(conserved therapy )

SUMMARY:
The objective of this study is to evaluate the therapeutic efficacy of allogenic bone marrow stem cells (BMSCs) transplantation in patients with liver cirrhosis. The evaluation of the efficacy includes the level of serum alanine aminotransferase (ALT), aspartate aminotransferase(AST), total bilirubin (TB),prothrombin time (PT), albumin (ALB), prealbumin(PA), precollagenⅢ(PCⅢ), collagenⅣ(Ⅳ-C), laminin(LN), hyaluronidase(HN), liver histological improvement before and 1 week to 1 year after transplantation. Child-Pugh scores and clinical symptoms were also observed simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16~65 years.
* Serum HBsAg positive for over six months.
* Ultrasonographic evidences of cirrhosis

Exclusion Criteria:

* History of moderate to severe hepatic encephalopathy or variceal bleeding during the last two months before enrolment.
* Prothrombin time is over 30s.
* Cirrhosis caused by other reasons except HBV infection.
* Severe problems in other vital organs(e.g.the heart,renal or lungs).
* Liver tumor on ultrasonography, CT or MRI examination.
* Pregnant or lactating women.
* Imaging evidences of vascular thromboses.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
Liver Function | 12 months

SECONDARY OUTCOMES:
Immunity | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lin B Liang, MD/PHD, Principal Investigator — SunYat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- See also: The Third Affiliated Hospital of Sun Yat-sen University — http://www.zssy.com.cn/